CLINICAL TRIAL: NCT03930199
Title: Personalized Mobility Interventions Using Smart Sensor Resources for Lower-Limb Prosthesis Users
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00208186
Record Dates: First submitted 2019-04-25; First posted 2019-04-29 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Amputation
Keywords: Prosthesis; Amputation; Prosthetic; Amputee; Smartphone; Sensors; Mobility
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Intervention Model Description: Upon enrollment, participants will be provided two sensors to track mobility and prosthesis use. Participants will wear the sensors continuously for 3 months and then will return to complete a set of assessments. The result of these assessments and analysis of sensor data will determine if the participant is meeting mobility goals and expected prosthesis use. Participants not meeting goals or prosthesis use will receive an intervention for 3 months. The intervention may include prosthetic care and physical therapy, or motivational interviewing, or both. During these 3 months, sensors will continue to monitor activity. After completion of intervention, participants will repeat the set of assessments and those who have improved in mobility goals and/or prosthesis use will continue to be monitored with sensors for an additional 3 months, after which the set of assessments will be completed a final time, assessing the maintenance of mobility goals and prosthesis use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Not Meeting Mobility Goals (Experimental): After the first three months of sensor monitoring, participants not meeting goals will receive an intervention (others will be removed from the study). The intervention assigned is not pre-determined, but will be assigned by an expert panel based on the individual needs determined from the assessment results and monitoring data. The intervention may include prosthetic care, physical therapy, motivational interviewing or other related psychological interventions, or a combination thereof. After three months of intervention, assessments are performed again and if improvement in prosthesis use is determined, participants are monitored for another three months to assess maintenance of prosthesis use (participants showing no improvement are removed from the study before these final three months of monitoring).
  Interventions: Other: Needs-based intervention (physical, psychological, or both)

INTERVENTIONS:
Other: Needs-based intervention (physical, psychological, or both) — Individuals identified as having physical issues (poor prosthesis fit, function, comfort or physical conditioning) will receive prosthetic care and physical therapy. This includes adjusting socket fit, component fit and repair, and in some instances replacement. Rehabilitation strategies include gait and prosthesis use retraining, balance fall-prevention, and range-of-motion training, strengthening, pain management, and activities of daily living training, based on participant-reported mobility goals. Individuals whose prosthesis use is reduced due to psychological issues will be provided with motivational interviewing and other related psychological interventions. During these interventions participant will be asked to set personal goals using a semi-structured interview that explores facilitators and barriers to wearing their prosthesis. If both physical and psychological issues are present, participant may receive both types of interventions simultaneously.

SUMMARY:
The goal of this research is to analyze data from smartphone-based and wearable sensors, using advanced machine-learning and data-mining techniques, and to combine this information with performance-based measures, participant-reported measures, and structured interviews to create a clinical toolbox to (i) identify individuals who exhibit reduced prosthesis use (compared to expected usage levels based on K-level designation and/or participant goals of community mobility and social interaction), (ii) identify prosthetic/physical and psychological factors that limit prosthesis use, and (iii) determine the effect of targeted interventions to increase prosthesis use and facilitate achievement of participant goals. Objective sensor-based measurement of home and community activities will allow for the correlation of real-world function to in-clinic assessments and to monitor changes resulting from rehabilitation interventions in real time. Machine-learning and data mining techniques will be used to identify a subset of measures from this toolbox that sensitively and accurately reflect real-world function, enabling clinicians to predict and assess activity and provide effective interventions to optimize prosthesis use. The goal of this project, to improve overall performance with respect to activities of daily living and other real-world activities, thus addresses the Fiscal Year 2017 (FY17) Orthotics and Prosthetics Outcomes Research Program (OPORP) Focus Area of Orthotic or Prosthetic Device Function.

DETAILED DESCRIPTION:
The overall goal of this research is to create a clinical toolkit to predict prosthesis use and function in the community. With this toolkit, clinicians will be able best determine an individual's K-Level designation, resulting in increased prosthesis use.

Aim 1: Determine whether a participant's prosthesis use matches the assigned K-level and/or self-reported goals and, if not, determine the reason(s) using an expert panel to evaluate data from performance-related measures, participant-reported measures, and smartphone and prosthesis sensors (clinical toolbox).

Aim 2: Quantify the effects of targeted physical intervention (prosthesis repair/refit, physical rehabilitation) or psychological intervention (motivational interviewing) or both on activity levels and patient goals.

Aim 3: Identify measure(s) that sensitively predict prosthesis use to create a clinically deployable toolkit to evaluate and optimize prosthesis use in the community.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral lower limb amputation at transtibial or transfemoral level
* Ability to wear and use a prosthesis
* Designated K-level 2 - 4, or equivalent
* Prescription of definitive prosthesis
* Veterans Affairs participants must receive care through the Veterans Affairs or related remote-site clinic
* Age: 18-89 years-to reflect the age range of eligible participants at Department of Defense and Veterans Affairs study sites, including young, combat-injured Service Members and healthy older Veterans, aged 70-80.

Exclusion Criteria:

* Co-morbidities that limit prosthesis use, independently of prosthetic function, training, or motivation, such as stroke, obesity, severe traumatic brain injury, and neuralgia, which require interventions outside the scope of this study. Suitability to participate in the study will be determined by the individual's physician.
* Unable or unwilling to learn to use the smartphone app or to allow transmission of study data
* Unable or unwilling to provide informed consent
* Residing in an area with poor cell phone coverage

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pre-intervention:10 Meter Walk Test (10MWT) | Week 12-13
  Assesses subject walking speed in meters per second for 10 meters. Subjects will repeat each measure 3 times at their normal self-selected walking speed and 3 times at a fast speed while still able to maintain safety.
Pre-intervention: 6 Minute Walk Test (6MWT) | Week 12-13
  The 6 minute walk test is performed as an objective evaluation of functional exercise capacity. The test measures the distance that the patient can walk on a flat, hard surface, indoors, in a period of 6 minutes. The walk test is patient self-paced and assesses the level of functional capacity. Patients are allowed to stop and rest during the test, however, the timer does not stop. If the patient is unable to complete the time, the time stopped is noted and reason for stopping prematurely is recorded.
Pre-intervention: Berg Balance Scale Test | Week 12-13
  This test is a standardized 14-item objective measure of postural stability and static balance; it is an established fall predictor in adults. Balance is measured during various tasks on a 5 point scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function, with a total possible score of 56. A score of 20 or less indicates a high fall risk.
Post-intervention:10 Meter Walk Test (10MWT) | Week 24-25
  Assesses subject walking speed in meters per second for 10 meters. Subjects will repeat each measure 3 times at their normal self-selected walking speed and 3 times at a fast speed while still able to maintain safety.
Post-intervention: 6 Minute Walk Test (6MWT) | Week 24-25
  The 6 minute walk test is performed as an objective evaluation of functional exercise capacity. The test measures the distance that the patient can walk on a flat, hard surface, indoors, in a period of 6 minutes. The walk test is patient self-paced and assesses the level of functional capacity. Patients are allowed to stop and rest during the test, however, the timer does not stop. If the patient is unable to complete the time, the time stopped is noted and reason for stopping prematurely is recorded. This test will be administered while wearing a mask to measure oxygen consumption.
Post-intervention: Berg Balance Scale Test | Week 24-25
  This test is a standardized 14-item objective measure of postural stability and static balance; it is an established fall predictor in adults. Balance is measured during various tasks on a 5 point scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function, with a total possible score of 56. A score of 20 or less indicates a high fall risk.
Delayed post-intervention:10 Meter Walk Test (10MWT) | Week 40-41
  Assesses subject walking speed in meters per second for 10 meters. Subjects will repeat each measure 3 times at their normal self-selected walking speed and 3 times at a fast speed while still able to maintain safety.
Delayed post-intervention: 6 Minute Walk Test (6MWT) | Week 40-41
  The 6 minute walk test is performed as an objective evaluation of functional exercise capacity. The test measures the distance that the patient can walk on a flat, hard surface, indoors, in a period of 6 minutes. The walk test is patient self-paced and assesses the level of functional capacity. Patients are allowed to stop and rest during the test, however, the timer does not stop. If the patient is unable to complete the time, the time stopped is noted and reason for stopping prematurely is recorded. This test will be administered while wearing a mask to measure oxygen consumption.
Delayed post-intervention: Berg Balance Scale Test | Week 40-41
  This test is a standardized 14-item objective measure of postural stability and static balance; it is an established fall predictor in adults. Balance is measured during various tasks on a 5 point scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function, with a total possible score of 56. A score of 20 or less indicates a high fall risk.

SECONDARY OUTCOMES:
Pre-intervention: Amputee Mobility Predictor (AMP) | Week 12-13
  The AMP is a tool used to predict the ambulatory potential of lower limb amputees, and measure function post-rehabilitation. It was developed to provide a more objective approach to rating amputees under the various K Classifications. The test can be performed with or without the prosthesis. The test involves activities of transfers, balance and walking. Score is out of 39 with each item scored in the range of 0-2.
Pre-intervention: Modified Falls Efficacy Scale (mFES) | Week 12-13
  The mFES is self-report questionnaire consisting of 14 items which is designed to measure fear of falling in the elderly. It assesses an individual's perception of balance during activities of daily living by asking "how confident are you that you can do the following activities without falling."
Post-intervention: Amputee Mobility Predictor (AMP) | Week 24-25
  The AMP is a tool used to predict the ambulatory potential of lower limb amputees, and measure function post-rehabilitation. It was developed to provide a more objective approach to rating amputees under the various K Classifications. The test can be performed with or without the prosthesis. The test involves activities of transfers, balance and walking. Score is out of 39 with each item scored in the range of 0-2.
Post-intervention: Modified Falls Efficacy Scale (mFES) | Week 24-25
  The mFES is self-report questionnaire consisting of 14 items which is designed to measure fear of falling in the elderly. It assesses an individual's perception of balance during activities of daily living by asking "how confident are you that you can do the following activities without falling."
Delayed post-intervention: Amputee Mobility Predictor (AMP) | Week 40-41
  The AMP is a tool used to predict the ambulatory potential of lower limb amputees, and measure function post-rehabilitation. It was developed to provide a more objective approach to rating amputees under the various K Classifications. The test can be performed with or without the prosthesis. The test involves activities of transfers, balance and walking. Score is out of 39 with each item scored in the range of 0-2.
Delayed post-intervention: Modified Falls Efficacy Scale (mFES) | Week 40-41
  The mFES is self-report questionnaire consisting of 14 items which is designed to measure fear of falling in the elderly. It assesses an individual's perception of balance during activities of daily living by asking "how confident are you that you can do the following activities without falling."

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (3):
- United States (3):
  - Shirley Ryan AbilityLab, Chicago, Illinois
  - Walter Reed National Military Medical Center, Center for Rehabilitation Sciences Research, Bethesda, Maryland
  - Minneapolis Veterans Affairs Health Care System, Minneapolis, Minnesota

REFERENCES:
- [Derived] B Aledi L, Flumignan CD, Trevisani VF, Miranda F Jr. Interventions for motor rehabilitation in people with transtibial amputation due to peripheral arterial disease or diabetes. Cochrane Database Syst Rev. 2023 Jun 5;6(6):CD013711. doi: 10.1002/14651858.CD013711.pub2. PMID 37276273

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT03930199/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT03930199/ICF_001.pdf